CLINICAL TRIAL: NCT04268589
Title: Effect of Virtual Reality Application on Pain, Functional Independence and Depression in Geriatric Individuals
Brief Title: Virtual Reality Effect in Geriatric Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Halil İbrahim Tuna, Director, Selcuk University
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: OGUU
Record Dates: First submitted 2020-01-21; First posted 2020-02-13 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Pain; Depression
Keywords: geriatric pain; geriatric depression
MeSH Terms: conditions — Pain; Depression

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): routine study
- virtual reality group (Experimental): Three days a week, 2 times a day, 15 minutes in the morning and in the evening for 9 days in total
  Interventions: Other: virtual reality game

INTERVENTIONS:
Other: virtual reality game — routine
  Other Names: routine
  Arms: virtual reality group

SUMMARY:
This study aimed to determine the effect of a virtual reality experience on pain, depression and functional adequacy in geriatric individuals living in a nursing home.

A virtual reality video with dance moves has been applied to the experimental group participants. Each video takes 3 minutes, and the elderly person has been put into practice at least 30 minutes after having breakfast in 3-minute periods and at least 30 minutes after dinner. In the morning and evening, 15 minutes, 2 times a day, a total of 9 days were applied for 3 weeks. The application lasted a total of 3 weeks. Scales were applied 1 week after the virtual reality application was completed and 1 month after the experimental group. The scales were filled in the control group at the same time.

DETAILED DESCRIPTION:
It is recommended that the future studies be conducted with larger samples on pain, depression, life quality and functionality.

ELIGIBILITY:
Inclusion Criteria:

* Suffering from musculoskeletal pain in the last 3 years,
* Being energetic (Being independent in the daily life activities),
* Being able to stand up without help before 30 seconds and walk at least six meters without help,
* Individuals with blood sugar ranging between 90-200 mg/dl prior to the application,
* Individuals with blood pressure ranging between 130-70 mm/Hg prior to the application,
* Not having neurological and psychiatric diseases,
* No history of fall,
* Being literate,
* Not being visually-hearing impaired,
* Being able to communicate verbally.

Exclusion Criteria:

* Pependent patients
* Patients with psychiatric illness
* Patients with joint pain disease diagnosis

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
The visual analog scale (VAS) | nine days
  This form includes numbers and is used in the assessment of pain severity. Patients mark their pain severity on a 10 cm ruler which is written no pain on one side and the most severe pain as possible on the other side. It has been stated that VAS is more sensitive and reliable in the measurement of pain severity than one sized scales
Geriatric Depression Scale | nine days
  The scale was developed by Yesavage with the aim of assessing the depression symptoms of old persons and consists of 15 questions in total. In the assessment, 1 point is given to each "no" answer in the positive questions and to each "yes" answer in the negative questions. A score of 6 and higher in the scale is accepted as meaningful for the diagnosis of depression. Reliability and validity tests were performed in our country and Chronbach alpha internal consistency coefficient was found to be 0.92

CONTACTS AND LOCATIONS:
Overall Officials: Gamze Unver, Principal Investigator — Kutahya University of Health Sciences; Halil Ibrahim Tuna, Principal Investigator — Selcuk University; Guler Balci Alparslan, Principal Investigator — Osmangazi University
Locations (1):
- Osmangazi University, Eskişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No